CLINICAL TRIAL: NCT06707155
Title: Study on the Use of Digital Platforms for the Control of Insulin Treatment in Patients With Type 1 Diabetes Mellitus
Brief Title: Digital Tracking With Auto Data Reporting
Status: Completed | Type: Observational
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: SUG_ART
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus (T1DM)
Keywords: T1DM; digital platforms; Remote patient monitoring; glycemic control; Caaring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Type 1 diabetes mellitus is a chronic pathology and represents a constant challenge for children and adolescents with diabetes and their families.

The objective of the treatment of DM1 in pediatric age is to achieve and maintain an optimal glycemic control in order to avoid or delay chronic micro- and macrovascular complications related to the disease.

However, currently, despite technological advances and the development of new insulin formulations, the majority of patients are unable to achieve glycemic goals.

In this context, the use of digital tools/platforms that allow remote monitoring of patients and that facilitate telemedicine have shown potential to improve treatment adherence and facilitate continued therapeutic education, improving clinical results with savings in time and associated costs.

DETAILED DESCRIPTION:
Patients are enrolled to a prospective, observational Post-Market clinical Follow-up study. This is a pilot study.

The protocol and informed consent documents have been reviewed and approved by the hospital human subjects reviewboard and the study will be performed in accordance with the Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients treated with subcutaneous insulin in multiple daily doses or patients treated with subcutaneous insulin in continuous subcutaneous infusion systems
* Patients using a glucose monitoring system
* Patients who are able to complete the study questionnaires
* Patients who are able to handle the application on a smart mobile phone.
* Informed consent is obtained from the patient.

Exclusion Criteria:

* Patients who, in the opinion of the investigator will not be able to commit to carrying out the follow-ups or do not have adequate technological skills

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from the Hospital Infantil Universitario Niño Jesús diagnosed with type 1 diabetes mellitus who meet the selection criteria and sign the informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Potential for improvement of type 1 diabetes through the use of a digital platform | 12 weeks
  Percentage of events related to diabetes reported through the use of a digital platform of the total events related to diabetes that occurred between medical visits.

SECONDARY OUTCOMES:
Degree of completion of data related to treatments between medical visits | Day 0 up to Week 12
  The Degree of completion of data related to treatments between medical is defined as the ratio between the questionnaires requested and completed.
Degree of completion of data related to intercurrent processes between visits | Day 0 up to Week 12
  The Degree of completion by patients of data related to intercurrent processes between is defined as the ratio between the questionnaires requested and completed
Degree of completion of therapeutic adherence between visits | Weekly up to 12 weeks
  The Degree of completion of therapeutic adherence by patients between visits is defined as the ratio between the questionnaires requested and completed.
Change in the patient's quality of life scale | Day 0 and week 12
  Change in the patient's quality of life scale the study compared to baseline. Health-Related Quality of Life in children and adolescents: Values (0-100), a higher score reflects a higher health-related quality of life (HRQoL).
Degree of completion of the questionnaires | Week 12
  Degree of completion of the questionnaires depending on age and gender, type of treatment and degree of glycemic control
Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIR | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIR (time in range)
Percentage of patients who complete the study correctly | Week 12
  Percentage of patients who complete the study correctly by completing all questionnaires
Variation in clinical parameters of glycemic control, HbA1c and CGM data: TBR | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: TBR (time below range)
Variation in clinical parameters of glycemic control, HbA1c and CGM data: CV | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: CV (Coefficient of Variation)
Variation in clinical parameters of glycemic control, HbA1c and CGM data: GRI | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: GRI (Glycemic Risk Index).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No